CLINICAL TRIAL: NCT06804746
Title: Safe Transplantation of Extended Criteria Donor Livers: Two-center Experience With Resuscitation and Viability Assessment of 206 Livers Using Sequential Hypo- and Normothermic Machine Perfusion
Brief Title: DCN for ECD Livers
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. Robert J. Porte, Head of HPB- and Transplant Surgery, Erasmus Medical Center
Other Study IDs: MEC-2024-0738
Record Dates: First submitted 2025-01-13; First posted 2025-02-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplantation
Keywords: Liver Transplantation; Machine Perfusion; Extended Criteria Donors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Adult patients (>18 years) who underwent liver transplantation of donor livers that required resuscitation and viability assessment through the previously published protocol for sequential hypo- and normothermic liver machine perfusion with controlled oxygenated rewarming (DHOPE-COR-NMP) based on a blood-based perfusate.
  Interventions: Procedure: DHOPE-COR-NMP

INTERVENTIONS:
Procedure: DHOPE-COR-NMP — Resuscitation and viability assessment through the previously published protocol of sequential hypo- and normothermic liver machine perfusion with controlled oxygenated rewarming (DHOPE-COR-NMP) based on a blood-based perfusate.

SUMMARY:
The goal of this observational study is to learn whether extended criteria donor livers can be safely transplanted after sequential hypo- and normothermic machine perfusion in recipients requiring a liver transplant for end-stage liver disease, including a long-term follow-up. The main questions it aims to answer are:

* Death censored graft-survival
* Overall patient survival
* Frequency of frequent post-transplant complications (e.g. non-anastomotic biliary strictures)

DETAILED DESCRIPTION:
With the increasing shortage of suitable donor livers for transplantation, extended criteria donor (ECD) livers may bridge the gap between available donor organs and donor livers needed. However, these ECD livers are associated with a higher risk of posttransplant complications. With the development of machine perfusion (MP) strategies over the recent years, (dual) hypothermic oxygenated perfusion ((D)HOPE) is established as a safe and effective way to reduce ischemia reperfusion injury. This leads to a decrease in early allograft dysfunction and non-anastomotic biliary strictures (NAS). On the other hand, normothermic machine perfusion (NMP) is mainly used for hepatobiliary functional assessment of liver grafts prior to transplantation. Combining both perfusion techniques through 1 hour of controlled oxygenated rewarming (COR), enables safe selection and transplantation of ECD livers after DHOPE-COR-NMP. Long-term outcomes are now available from two centers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Donor livers that required resuscitation and viability assessment through the previously published sequential hypo- and normothermic liver machine perfusion (DHOPE-COR-NMP) protocol based on a blood-based perfusate.

Exclusion Criteria:

* Multiorgan transplantation
* Split liver transplant
* Living donor liver transplantation
* Previous donor organ perfusion (e.g. Normothermic Regional Perfusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years) undergoing liver transplantation of extended criteria donor livers, which therefore required resuscitation and viability assessment through the previously published DHOPE-COR-NMP protocol based on a blood-based perfusate.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Death-censored graft survival | 1 year post-transplant
  Time from liver transplantation until re-transplantation or death due to graft dysfunction, with censoring of subjects who died with a functioning graft.

SECONDARY OUTCOMES:
Overall patient survival | 1 year post-transplant
  Time from liver transplantation until all-cause death
• Overall graft survival | 1 year post-transplant
  Time from liver transplantation until re-transplantation or all-cause death.
Number of participants with primary non function | From transplantation until 7 days post-transplant
  Livers failing to sustain their primary function, leading to death or re-transplantation within 7 days of the primary procedure, in the presence of patent blood supply and outflow (8).
Occurrence of hepatic arterial thrombosis | 1 year post-transplant
  Radiologically or surgically proven thrombosis of the hepatic artery.
Occurrence of portal vein thrombosis | 1 year post-transplant
  Radiologically or surgically proven thrombosis of the portal vein.
Occurrence of venous outflow tract obstruction | 1 year post-transplant
  Radiologically or surgically proven thrombosis of the main hepatic veins or the inferior vena cava.
Occurrence of non-anastomotic biliary strictures | 1 year post-transplant
  Any irregularity or narrowing of the lumen of the intrahepatic or extrahepatic donor bile ducts, excluding the biliary anastomosis, diagnosed with the use of cholangiography in combination with clinical symptoms (e.g., jaundice or cholangitis) or an elevation of cholestatic laboratory variables, in the presence of a patent hepatic artery (5).
Occurrence of anastomotic biliary strictures | 1 year post-transplant
  Strictures occurring at the anastomosis of donor choledochal duct and recipient choledochal duct or jejunal Roux-limb.
Occurrence of biliary leakage | From 3 days after transplantation until the the first year post-transplant
  Fluid with an elevated (>3x serum) bilirubin level in the abdominal drain or intra-abdominal fluid on or after post-operative day 3 or the need for radiological intervention (i.e. interventional drainage) owing to biliary collections or re-laparotomy due to biliary peritonitis (9).
Biliary complications: as a composite | 1 year post-transplant
  A composite of individually studied outcome measures (reported as one single outcome measure), composed of: non-anastomotic biliary strictures, anastomotic biliary strictures and biliary leakage.
Intensive care stay | From transplantation until discharge from the Intensive care unit to the ward after transplantation or date of death from any cause during initial admission, whichever came first, assessed up to 6 months
  Intensive care stay post-transplantation
Total hospital stay | From transplantation until discharge after transplantation, or date of death from any cause during initial admission, whichever came first, assessed up to 6 months
  Defined as total hospital stay from transplantation until discharge, including intensive care unit stay

OTHER OUTCOMES:
Composite of post-transplant incidence of biliary interventions | Until 6 months after liver transplantation
  The occurrence and frequency of the composite of one of the following biliary interventions (reported as one single outcome measure): Endoscopic Retrograde Cholangio- and Pancreaticography, drainage performed by percutaneous transhepatic cholangiography and re-interventions for biliary complications (e.g. bile leaks)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Erasmus Medical Center, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Vries Y, Berendsen TA, Fujiyoshi M, van den Berg AP, Blokzijl H, de Boer MT, van der Heide F, de Kleine RHJ, van Leeuwen OB, Matton APM, Werner MJM, Lisman T, de Meijer VE, Porte R. Transplantation of high-risk donor livers after resuscitation and viability assessment using a combined protocol of oxygenated hypothermic, rewarming and normothermic machine perfusion: study protocol for a prospective, single-arm study (DHOPE-COR-NMP trial). BMJ Open. 2019 Aug 15;9(8):e028596. doi: 10.1136/bmjopen-2018-028596. PMID 31420387
- [Background] van Leeuwen OB, de Vries Y, Fujiyoshi M, Nijsten MWN, Ubbink R, Pelgrim GJ, Werner MJM, Reyntjens KMEM, van den Berg AP, de Boer MT, de Kleine RHJ, Lisman T, de Meijer VE, Porte RJ. Transplantation of High-risk Donor Livers After Ex Situ Resuscitation and Assessment Using Combined Hypo- and Normothermic Machine Perfusion: A Prospective Clinical Trial. Ann Surg. 2019 Nov;270(5):906-914. doi: 10.1097/SLA.0000000000003540. PMID 31633615
- [Background] van Rijn R, Schurink IJ, de Vries Y, van den Berg AP, Cortes Cerisuelo M, Darwish Murad S, Erdmann JI, Gilbo N, de Haas RJ, Heaton N, van Hoek B, Huurman VAL, Jochmans I, van Leeuwen OB, de Meijer VE, Monbaliu D, Polak WG, Slangen JJG, Troisi RI, Vanlander A, de Jonge J, Porte RJ; DHOPE-DCD Trial Investigators. Hypothermic Machine Perfusion in Liver Transplantation - A Randomized Trial. N Engl J Med. 2021 Apr 15;384(15):1391-1401. doi: 10.1056/NEJMoa2031532. Epub 2021 Feb 24. PMID 33626248
- [Background] Eden J, Bruggenwirth IMA, Berlakovich G, Buchholz BM, Botea F, Camagni S, Cescon M, Cillo U, Colli F, Compagnon P, De Carlis LG, De Carlis R, Di Benedetto F, Dingfelder J, Diogo D, Dondossola D, Drefs M, Fronek J, Germinario G, Gringeri E, Gyori G, Kocik M, Kucukerbil EH, Koliogiannis D, Lam HD, Lurje G, Magistri P, Monbaliu D, Moumni ME, Patrono D, Polak WG, Ravaioli M, Rayar M, Romagnoli R, Sorensen G, Uluk D, Schlegel A, Porte RJ, Dutkowski P, de Meijer VE. Long-term outcomes after hypothermic oxygenated machine perfusion and transplantation of 1,202 donor livers in a real-world setting (HOPE-REAL study). J Hepatol. 2025 Jan;82(1):97-106. doi: 10.1016/j.jhep.2024.06.035. Epub 2024 Jul 3. PMID 38969242
- [Background] Schlegel A, Porte R, Dutkowski P. Protective mechanisms and current clinical evidence of hypothermic oxygenated machine perfusion (HOPE) in preventing post-transplant cholangiopathy. J Hepatol. 2022 Jun;76(6):1330-1347. doi: 10.1016/j.jhep.2022.01.024. PMID 35589254
- [Background] Foley DP, Fernandez LA, Leverson G, Anderson M, Mezrich J, Sollinger HW, D'Alessandro A. Biliary complications after liver transplantation from donation after cardiac death donors: an analysis of risk factors and long-term outcomes from a single center. Ann Surg. 2011 Apr;253(4):817-25. doi: 10.1097/SLA.0b013e3182104784. PMID 21475025
- [Background] Nemes B, Gaman G, Polak WG, Gelley F, Hara T, Ono S, Baimakhanov Z, Piros L, Eguchi S. Extended-criteria donors in liver transplantation Part II: reviewing the impact of extended-criteria donors on the complications and outcomes of liver transplantation. Expert Rev Gastroenterol Hepatol. 2016 Jul;10(7):841-59. doi: 10.1586/17474124.2016.1149062. Epub 2016 Mar 2. PMID 26831547